CLINICAL TRIAL: NCT06734026
Title: Multimodal, Enriched Environment for Rehabilitation
Brief Title: Multimodal, Enriched Environment for Rehabilitation in Chronic Traumatic Brain Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, James Sulzer, Principal Investigator, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Study00000332; HD116036 (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2024-12-05; First posted 2024-12-13 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2024-11

CONDITIONS: Traumatic Brain Injury (TBI) Patients
Keywords: TBI; Brain injury; Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cafe Therapy (Experimental): Participants will be volunteer workers for two hours per day, three days per week for 6-8 weeks, alongside a trained researcher.
  Interventions: Behavioral: Cafe Therapy
- Control Group (No Intervention): No Intervention is administered during the 2 months between Assessments

INTERVENTIONS:
Behavioral: Cafe Therapy — Participants will be volunteer workers for two hours per day, three days per week for 6-8 weeks, alongside a trained researcher. Participants will complete at least 18 sessions of training within the time frame. Participants will run the Café with supervision from a researcher, serving customers prepackaged food and drinks per our protocol, along with guidance and direction from a therapist, once a week. Participants will be responsible for interacting with customers and arranging supplies. On a weekly basis, participants will be asked how they feel (for example tired, stressed, overwhelmed, etc) before and after their session and to rate how well they performed in the café.
  Arms: Cafe Therapy

SUMMARY:
The goal of this study is to learn if a enhanced environment (Metro Café) with multi model approach (an approach that combines several therapies) in chronic traumatic brain injury improves outcomes of recovery better than traditional therapy. The main questions it aims to answer are:

* Determine the amount of therapy dosage (speech, cognition, arm and leg movements) obtained during the Metro Café therapy session.
* Evaluate the connection between environmental enrichment dosage (the Metro Café) and clinical outcome scores.

Researchers will compare Metro Café Treatment to those who do not receive this treatment to see if better improvements in function after a traumatic brain injury are seen in the Metro Café Treatment Participants will train in the Metro Cafe during the 2-month gap between assessments, for a total of 18 training sessions, each up to 2 hours, 3 times per week. Participants will greet and serve customers drinks and snacks, maintain food supplies at the counters and performs housekeeping tasks with advice and assistance from a supervising researcher as needed,

DETAILED DESCRIPTION:
People who have had a brain injury and their caregiver, are being asked to participate in this study. After a brain injury it is a common to have cognitive and physical limitations. These problems can lead to the inability to care for yourself, lack of motivation, isolation, and loss of employment. Therapies are commonly prescribed to address these issues. The standard of care is to prescribe physical, occupational and speech therapy. If you are thinking about this study, you have probably tried some of these treatments. Therapies typically address walking, balance, reaching and grasping as well as problem-solving and memory, with the goal to complete as many repetitions of the activities as possible to improve your overall function. However, this therapy does not always address real life activities.

We have developed an enhanced environment for multimodal therapy called "The Metro Café." This is a free-standing frame on an adjustable body weight support system which allows you to move in a small area. The harness wraps around your torso and is attached to an overhead frame to prevent falls and reduce some of your weight making mobility easier. Participants in this portion of the study will operate a small Café serving food and drinks. The goal of this therapy is for participants to practice job activities that involve motor, social and cognitive skills.

The purpose of this study is to determine if a multimodal approach (an approach that combines several different therapies) to therapy results in improved outcomes for recovery after a brain injury.

Participants assigned to the Metro Cafe treatment will work in a cafe setting 3x/week for 2 months. Participants will greet and serve customers drinks and snacks, maintain food supplies at the counters and performs housekeeping tasks with advice and assistance from a supervising researcher as needed.

Some participants will not receive treatment and will only complete the study Assessments.

Participants and Caregiver will complete Survey before and after the treatment. Participants will also complete functional assessments of Upper and Lower extremity function, gait and balance.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe neurological diagnosis as diagnosed by a clinician,
* ability to comprehend multi step instructions,
* ability to independently balance with weight support,
* physical deficits resulting in need for additional functional goals,
* ability to endure 2 hours of weight-supported standing,
* ability to provide informed consent,
* basic communication ability,
* currently discharged from therapy,
* >3 months post-injury,
* >18 years of age at time of enrollment

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Non-English speaking
* Pregnant women
* Prisoners
* Medical instability
* Other neurological conditions
* Severe problems with maintaining follow-up expected (such as, but not limited to history of substance abuse, homelessness/incarceration, dementia and psychotic disorders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2028-01-15 (Estimated); Study Completion 2029-01-15 (Estimated)

PRIMARY OUTCOMES:
Limb Motion Analysis | Baseline, 10 weeks post treatment
  Preprocessing of data will be performed, and motion data will then be extracted. We will evaluate motion by single limb, namely: right arm, right leg, left arm, left leg. We will also combine across limbs: right arm, left arm, right leg, left leg, and over the whole-body amount of motion (AoM).

SECONDARY OUTCOMES:
10 Meter Walk Test (10-MWT) | Baseline, 10 weeks post treatment
  The total time taken to ambulate 6 meters (m) is recorded to the nearest hundredth of a second. 6 m is then divided by the total time (in seconds) taken to ambulate and recorded in m/seconds
Action Research Arm Test (ARAT) | Baseline, 10 weeks post treatment
  The Action Research Arm Test (ARAT) is a 19-item measure aimed at assessing functional performance of the upper extremity through observational means.
Neuro - Qol(Quality of Life) | Baseline, 10 weeks post treatment
  The NeuroQOL is a self-report of health related quality of life in 17 domains and sub-domains for adults and 11 for children with neurological disorders. The measure is available for administration via Computer Assisted Testing or in short forms (8-10 items) for each sub-domain that can be selected based on individual patient needs:
  * Neuro-QoL - Positive Affect and Well-Being the following Domains will be used:
  * Neuro-QoL - Lower Extremity Function
  * Neuro-QoL - Upper Extremity Function
  * Neuro-QoL - Sleep Disturbance
  * Neuro-QoL - Emotional and Behavioral Dyscontrol
  * Neuro-QoL - Fatigue
  * Neuro-QoL - Stigma
  Scale 1-5 (lower score better outcome)
  1. - Never
  2. - Rarely
  3. - Sometimes
  4. - Often
  5. - Always

CONTACTS AND LOCATIONS:
Overall Officials: James Sulzer, PhD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make the IPD available.